CLINICAL TRIAL: NCT01215695
Title: Feasibility of a Combined Use of a Video-laryngoscope With a Novel Video-stylet for Predicted Difficult Intubation
Brief Title: Video-laryngoscope With a Novel Video-stylet for Difficult Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rainer Lenhardt, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UofL IRB #10.0300
Record Dates: First submitted 2010-07-22; First posted 2010-10-06 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Difficult Endotracheal Intubation
Keywords: Intubation, Endotracheal; Endotracheal Intubation, adverse events

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients will be randomly assigned to having their ETT placed with use of a pre-formed stylet provided by the manufacturer of the GVL (control group)
  Interventions: Device: Control
- Intervention (Experimental): Patients will be randomly assigned to either having their ETT placed with use of flexible, disposable tracheoscope (aScope, Ambu, Denmark) (intervention group).
  Interventions: Device: aScope (Ambu Inc. 6740 Baymeadow Drive Glen Burnie, MD)

INTERVENTIONS:
Device: aScope (Ambu Inc. 6740 Baymeadow Drive Glen Burnie, MD) — The aScope is a flexible, disposable plastic tracheoscope that incorporates a high-resolution video camera with an LED light at its flexible tip and has attached monitor.
  Other Names: video-stylet
  Arms: Intervention
Device: Control — pre-formed stylet provided by the manufacturer of the GlideScope® video laryngoscope
  Arms: Control

SUMMARY:
We propose to enroll 140 subjects scheduled for elective or urgent/emergent surgery with general anesthesia including endotracheal intubation. Patients qualify for the trial if they are considered a difficult airway case as determined by measurement of common predictive indices for difficult intubation (see inclusion criteria). All patients will be intubated with a GVL. Patients will be randomly assigned to either having their ETT placed with use of a pre-formed stylet provided by the manufacturer of the GVL (control group) or with a flexible, disposable tracheoscope (aScope, Ambu, Denmark) (intervention group). The randomization will be stratified as to whether patients are categorized as predicted difficult airway or have an immobilized cervical spine (C-collar in place).

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* Thyromental distance < 6 cm
* Sterno-mental distance < 12 cm
* Mallampati grade 3 and 4
* Interincisor distance < 38 mm
* Status of dentition: presence of buckteeth
* Neck movement < 35°
* Neck circumference >43 cm at the level of the thyroid cartilage
* Patients with immobilized cervical spine (C-collar in place).
* History of difficult laryngoscopy or intubation

Exclusion Criteria:

* Full stomach
* Hiatal hernia
* Severe GERD (Gastroesophageal reflux disease)
* Tumors of the upper airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Lenhardt, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Result] Lenhardt R, Burkhart MT, Brock GN, Kanchi-Kandadai S, Sharma R, Akca O. Is video laryngoscope-assisted flexible tracheoscope intubation feasible for patients with predicted difficult airway? A prospective, randomized clinical trial. Anesth Analg. 2014 Jun;118(6):1259-65. doi: 10.1213/ANE.0000000000000220. PMID 24842175

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 46 (14) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 27 | 64
  Male | 33 | 43 | 76
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time
Description: divided into time to successfully place the glidescope (visualization of the epiglottis), time to successfully insert the videostylet (passing through the cords) and time to verified placement of the ETT (as outlined above). Interim bag and mask time, if needed, will not be included in the intubation time. More than 5 attempts or 120 s are regarded as failure of intubation. If failure to secure the airway occurs with the GVL and videostylet, then conventional difficult intubation protocols approved by the University of Louisville Hospital will be implemented.
Time Frame: 120 seconds
Measure: Median (Inter-Quartile Range); unit: time in seconds
Arm/Group | Control | Intervention
Number analyzed (Participants) | 70 | 70
time in seconds | 66 [47 to 89] | 71 [52 to 100]
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Number of Intubation Attempts
Description: counted as each approach of the ETT to the glottic entrance.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Number of intubation attempts
Arm/Group | Control | Intervention
Number analyzed (Participants) | 70 | 70
Number of intubation attempts | 1.2 (0.6) | 1.1 (0.4)
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Neck Movement
Description: One observer will video-record the entire intubation procedure. At a later time, an otherwise unrelated observer will watch the video-records and grade the neck movement during intubation. Neck movement will be classified as Grade 0: no neck movement, Grade 1: minimal neck movement, or Grade 2: moderate neck movement. Results are reported as total with mild, moderate, or severe neck movement.
Time Frame: 30 minutes
Population: Only those participants with available data were analyzed for the assessment. All subjects reported had mild, moderate or severe neck movement.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 47 | 54
Participants | 47 | 54
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.05, Chi-squared

4. Secondary Outcome: Laryngeal View Grade of 1 or 2
Description: The laryngeal view as Grade 1 (full view of the glottis) or Grade 2 (glottis partly exposed, anterior commissure not seen) according to the method described by Cormack and Lehane (1984).
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 70 | 70
Participants | 62 | 50
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.05, Chi-squared

5. Secondary Outcome: Ease of Intubation
Description: After completion of the procedure the intubator will be asked to score the ease of intubation. To do this, he/she will give a score from 0-100 with 0 being the easiest and 100 being the hardest.
Time Frame: 2-4 hours after intubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 70 | 70
units on a scale | 36 (23) | 39 (25)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/70 | 2/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=70) | Intervention (N=70)
Unable to intubate (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — Four patients could not be intubated with VLS and rigid stylet. These patients were subsequently intubated successfully using the alternative method with a complementary flexible tracheoscope

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes